CLINICAL TRIAL: NCT01435512
Title: Strength At Home: Veterans' Program (Formerly: Post-Traumatic Stress Disorder (PTSD)-Focused Therapy for Anger and Relationship Conflict Among Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans)
Brief Title: Strength At Home: Veterans' Program (PTSD-Focused Therapy for Anger and Relationship Conflict Among OEF/OIF Veterans)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Casey Taft, Principal Investigator, Boston VA Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT073945
Record Dates: First submitted 2009-08-06; First posted 2011-09-16 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Domestic Violence
Keywords: PTSD; CBT; Intimate Partner Violence; Treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group (Experimental): PTSD-Focused Cognitive Behavioral Therapy for Partner Violence
  Interventions: Behavioral: PTSD-Focused CBT for Partner Violence
- Waitlist (No Intervention): Control group - no intervention

INTERVENTIONS:
Behavioral: PTSD-Focused CBT for Partner Violence — PTSD-Focused CBT (PFCBT) will consist of 12 2-hour weekly sessions,led by two project therapists. In each session, group members will discuss materials and do assignments to practice skills.
  Other Names: Strength at Home; Veterans Program
  Arms: Group

SUMMARY:
This is a research study funded by the Department of Defense to test a therapeutic intervention for male combat veterans who engage in intimate partner violence (IPV). The investigators hope to decrease the recurrence of relationship aggression and help veterans manage anger. The primary aim of the study is to test the intervention.

DETAILED DESCRIPTION:
The purpose of this project is to develop, standardize, and test an intervention for combat veterans exposed to trauma who engage in intimate partner aggression (IPA). This intervention, formerly labeled PTSD-Focused Cognitive Behavior Therapy for Partner Violence (PFCBT), and currently called the Strength at Home, Veteran's Program, incorporates components of interventions for IPA and trauma and will target mechanisms implicated in the relationship between trauma and IPA. This project addresses a number of the research gaps in this area of research including: (a) the development of a novel treatment approach to improve functioning and well-being of affected individuals; (b) tertiary prevention (of repeated IPA) during re-integration; and (c) examination of the efficacy of a program providing support for the families and caregivers of veterans with combat history.

ELIGIBILITY:
Inclusion Criteria:

* Any era veteran
* Over the age of 18
* In a relationship within a female partner within the last 6 months
* At least one act of male-to-female physical aggression over the previous 6 months or at least one act of male-to-female severe violence in the past 12 months
* Male participant must consent for partner contact

Exclusion Criteria:

* Participant evidences severe organicity or active psychosis
* Reading difficulties prevent valid completion of the assessment instruments
* Participant expresses prominent suicidal or homicidal ideation
* Participant meets diagnostic criteria for alcohol and/or drug dependence, if not in early full remission or sustained partial remission

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2009-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Casey T. Taft, PhD, Principal Investigator — VA Boston Healthcare System; Suzannah Creech, PhD, Principal Investigator — VA VISN 17 Center of Excellence
Locations (2):
- United States (2):
  - National Center for PTSD/VA Boston Healthcare System, Boston, Massachusetts
  - Providence VA Medical Center, Providence, Rhode Island

REFERENCES:
- [Result] Taft CT, Macdonald A, Creech SK, Monson CM, Murphy CM. A Randomized Controlled Clinical Trial of the Strength at Home Men's Program for Partner Violence in Military Veterans. J Clin Psychiatry. 2016 Sep;77(9):1168-1175. doi: 10.4088/JCP.15m10020. PMID 26613288
- [Derived] Creech SK, Macdonald A, Benzer JK, Poole GM, Murphy CM, Taft CT. PTSD symptoms predict outcome in trauma-informed treatment of intimate partner aggression. J Consult Clin Psychol. 2017 Oct;85(10):966-974. doi: 10.1037/ccp0000228. Epub 2017 Jul 20. PMID 28726440
- See also: Taft CT, Macdonald A, Creech SK, Monson CM, Murphy CM. A randomized controlled clinical trial of the Strength at Home Men's Program for partner violence in military veterans. J Clin Psychiatry. 2015 Nov 24. [Epub ahead of print] — http://dx.doi.org/10.4088/JCP.15m10020

RESULTS

PARTICIPANT FLOW:
Groups:
- PTSD-Focused Cognitive Behavioral Therapy for Partner Violence: PTSD-Focused Cognitive Behavioral Therapy for Partner Violence
  PTSD-Focused CBT for Partner Violence: PTSD-Focused CBT (PFCBT) will consist of 12 2-hour weekly sessions,led by two project therapists. In each session, group members will discuss materials and do assignments to practice skills.
- Waitlist: Control group - no intervention. Participants who were randomized to the waitlist at baseline were offered PTSD-Focused Cognitive Behavioral Therapy for Partner Violence after the 3-month follow-up.
Period: Overall Study
Arm/Group | PTSD-Focused Cognitive Behavioral Therapy for Partner Violence | Waitlist
Started | 67 | 68
Completed | 67 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group | Waitlist | Total
Number analyzed (Participants) | 67 | 68 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 68 | 135
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (12.9) | 38.2 (12.7) | 37.85 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 67 | 68 | 135
Region of Enrollment [Number; unit: participants]
  United States | 67 | 68 | 135

OUTCOME MEASURES:

1. Primary Outcome: Intimate Partner Aggression as Measured by the Conflict Tactics Scale
Description: Revised Conflict Tactics Scale-2 (CTS2). The CTS2 is the most widely used measure of IPV, with excellent internal consistency reliability, content validity, and construct validity.76,88 Combined partner reports will be used such that scores of partners who report a greater frequency of specific CTS2 behaviors will be used in analyses to reduce the impact of response biases and the underreporting of abuse. The CTS2 will also be given every four weeks during the course of active intervention. Scale response options range from 0 to 7. Higher overall scores mean more conflict.
Time Frame: Pretreatment (baseline), Posttreatment (12 weeks), 3 month follow up (24 weeks)
Measure: Mean (95% Confidence Interval); unit: Mean CTS Score
Arm/Group | Group | Waitlist
Number analyzed (Participants) | 67 | 68
Mean CTS Score
  Pretreatment Physical IPV | 2.82 [2.19 to 3.45] | 2.51 [1.9 to 3.13]
  Posttreatment Physical IPV | 0.71 [0.33 to 1.1] | 1.69 [1.01 to 2.38]
  Follow up Physical IPV | 0.80 [0.18 to 1.41] | 0.80 [0.37 to 1.23]
  Pretreatment Psychological IPV | 4.43 [3.87 to 5.0] | 4.46 [3.94 to 4.99]
  Posttreatment Psychological IPV | 2.81 [2.21 to 3.41] | 3.87 [3.2 to 4.54]
  Follow up Psychological IPV | 3.04 [2.35 to 3.73] | 3.69 [3.11 to 4.26]

2. Secondary Outcome: Multidimensional Measure of Emotional Abuse (MMEA)
Description: Change of physical and psychological IPV as evidenced by reduction in MMEA scores. MMEA is a 28-item measurement tool with scale responses ranging from 0 to 7 where higher scores indicate greater emotional abuse.
Time Frame: Pretreatment (baseline), Posttreatment (12 weeks), 3 month follow up (24 weeks)
Measure: Mean (95% Confidence Interval); unit: MMEA Scores
Arm/Group | Group | Waitlist
Number analyzed (Participants) | 67 | 68
MMEA Scores
  MMEA Restrictive Engulfment Pretreatment | 3.47 [2.89 to 4.05] | 3.93 [3.40 to 4.45]
  MMEA Restrictive Engulfment Posttreatment | 2.11 [1.54 to 2.68] | 3.35 [2.73 to 3.97]
  MMEA Restrictive Engulfment Follow Up | 1.80 [1.21 to 2.38] | 3.24 [2.61 to 3.86]
  MMEA Denigration Pretreatment | 3.21 [2.66 to 3.76] | 3.49 [2.9 to 4.07]
  MMEA Denigration Posttreatment | 1.80 [1.23 to 2.36] | 2.82 [2.19 to 3.45]
  MMEA Denigration Followup | 2.35 [1.68 to 3.02] | 2.51 [1.89 to 3.13]
  MMEA Hostile Withdrawal Pretreatment | 5.63 [5.14 to 6.12] | 5.84 [5.38 to 6.29]
  MMEA Hostile Withdrawal Posttreatment | 4.1 [3.39 to 4.82] | 4.95 [4.24 to 5.65]
  MMEA Hostile Withdrawal Follow up | 3.94 [3.22 to 4.67] | 5.03 [4.41 to 5.66]
  MMEA Dominance/Intimidation Pretreatment | 3.79 [3.22 to 4.37] | 3.46 [2.89 to 4.02]
  MMEA Dominance/Intimidation Posttreatment | 2.20 [1.61 to 2.79] | 2.64 [2.01 to 3.27]
  MMEA Dominance/Intimidation Followup | 1.91 [1.29 to 2.53] | 1.92 [1.37 to 2.46]

3. Secondary Outcome: Symptoms of Posttraumatic Stress Disorder as Assessed by the Clinician Administered PTSD Scale (CAPS) and the Posttraumatic Stress Disorder Checklist (PCL)
Description: PTSD was used as a predictor instead of an outcome measure to determine if PTSD status was associated with poorer treatment response compared to the treatment as usual group. Refer to Creech and colleagues (2017). The structured interview utilizing CAPS was used to assess the frequency and intensity of the PTSD symptoms. Response options range from 1 "Not at all" to 5 "Extremely" for a total symptom severity score range of 17-85. Higher scores indicate symptoms severity of PTSD.
  Creech, S. K., Macdonald, A., Benzer, J. K., Poole, G. M., Murphy, C. M., & Taft, C. T. (2017, July 20). PTSD Symptoms Predict Outcome in Trauma-Informed Treatment of Intimate Partner Aggression. Journal of Consulting and Clinical Psychology. http://dx.doi.org/10.1037/ccp0000228
Time Frame: 6 month follow-up (72 weeks)
Reporting Status: Not Posted

4. Secondary Outcome: Relationship Satisfaction as Measured by the Dyadic Adjustment Scale
Description: Changes in relationship satisfaction as evidenced by answers to the Dyadic Adjustment Scale. Items 1-15 options: Always Agree, Almost Always Agree, Occasionally Disagree, Frequently Disagree, Almost Always Disagree, Always Disagree. Item 16-22: All the Time, Most of the Time, More Often than Not, Rarely, Never. Item 23: Every day, Almost Every Day, Occasionally, Rarely, Never. Item 24: All of them, Most of them, Some of them, Very few of them, None of them. Items 25-28: Never, Less than once a month, Once or twice a month, Once or twice a week, Once a day, More often. Items 29-30: Yes/No. Item 31: Extremely Unhappy, Fairly Unhappy, A Little Unhappy, Happy, Very Happy, Extremely Happy, Perfect. Item 32: six statements in which the participant picks the statement that best describes how they feel about the future of their relationship. Overall score ranges from 0 to 151; higher scores indicating a more positive adjustment and lower level of distress within relationship.
Time Frame: 6-month follow up (72 weeks)
Reporting Status: Not Posted

5. Secondary Outcome: Trait Anger as Measured by the State-Trait Anger Expression Inventory (STAXI) and Aggression as Measured by the Aggression Questionnaire
Description: 57 items assessing the intensity of anger as an emotional state (State Anger) and the tendency of an individual to experience state anger, or anger proneness (Trait Anger).
  The Trait Anger scale measures individual differences in the disposition to experience anger. The Anger Expression scale provides an index of the frequency of anger expression. Response options are 1 (not at all/hardly ever), 2 (somewhat/sometimes), or 3 (Very Much/Often). There are several subscales and, in general, higher scores indicate great feelings of anger, more likely to express anger, etc.
Time Frame: 6-month follow up (72 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- PTSD-Focused Cognitive Behavioral Therapy Group: PTSD-Focused Cognitive Behavioral Therapy for Partner Violence
  PTSD-Focused CBT for Partner Violence: PTSD-Focused CBT (PFCBT) will consist of 12 2-hour weekly sessions,led by two project therapists. In each session, group members will discuss materials and do assignments to practice skills.
- Control Group: Control Group
  Control Group: The study utilized a wait list control. Individuals on the wait list did not receive an intervention.
Arm/Group | PTSD-Focused Cognitive Behavioral Therapy Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/68
Other Adverse Events (participants affected / at risk) | 0/67 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No